CLINICAL TRIAL: NCT01457482
Title: Art Therapy as Treatment for Fear of Childbirth:a Randomized Controlled Study
Brief Title: Art Therapy as Treatment for Fear of Childbirth
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Helsingborgs Hospital (Other)
Responsible Party: Principal Investigator, Helen Wahlbeck, Lic.Midwife, Art therapist, Helsingborgs Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 210/422
Record Dates: First submitted 2011-10-19; First posted 2011-10-24 (Estimated); Last update posted 2012-02-14 (Estimated); Status verified 2012-02

CONDITIONS: Fear of Childbirth
Keywords: Fear; Childbirth; Art therapy; Therapeutic conversations; W-DEQ
MeSH Terms: interventions — Art Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Art therapy group (Experimental): Treatment in this arm consists of five Art Therapy sessions and therapeutic conversations.
  Interventions: Other: Art Therapy and therapeutic conversations
- Therapeutic conversation group (Active Comparator): Treatment by therapeutic conversations only
  Interventions: Other: Therapeutic conversations

INTERVENTIONS:
Other: Art Therapy and therapeutic conversations — Treatment consists of five sessions of Art Therapy given by an authorised Art Therapist and therapeutic conversations with specialist midwives. Number of conversations is determined by the participant.
  Arms: Art therapy group
Other: Therapeutic conversations — Therapeutic conversations with specialist midwives. Number of conversations is determined by the participant.
  Arms: Therapeutic conversation group

SUMMARY:
Earlier research has shown that pregnant women with a pronounced fear of childbirth have a significantly increased risk for birth complications and subsequent psychological trauma. In Sweden and also internationally, women in fear of childbirth are treated in many differing ways. Evidence for best care for these women is lacking. The Art Therapy method is a creative, psycho-therapeutic form of treatment which has been used for several decades within psychiatry. It has recently been seen that the Art Therapy method has positive effects during treatment for crisis reactions.

Recruitment has recently been initiated for a randomized controlled study of Art Therapy for the treatment of fear of childbirth.

The hypothesis for the study is as follows:

H1 = treatment with Art Therapy and therapeutic conversations will result in a decrease in fear of childbirth when compared to treatment by therapeutic conversations only.

The instrument which is to be used for measurement of childbirth fear is the Wijma Delivery Expectancy Questionnaire (W-DEQ). This is a well validated instrument which was developed in Sweden. A power calculation has shown a need for 62 x 2 participants; a total of 124 women.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women
* Pronounced fear of childbirth

Exclusion Criteria:

* Women with a current psychiatric diagnosis
* Women who do not understand Swedish
* Women with a current substance misuse

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 124 (Estimated)
Dates: Start 2011-05; Primary Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Scores for the Wijma Delivery Expectancy Questionnaire (W-DEQ) | Change in W-DEQ scores measured at entry to the study (approximately gestational weeks 20 to 31) and again at gestational week 36.

CONTACTS AND LOCATIONS:
Overall Officials: Linda J Kvist, PhD, Study Chair — Lund University, Lund, Sweden
Locations (1):
- Helsingborg Hospital, Helsingborg, Skåne County, Sweden

REFERENCES:
- [Derived] O'Connell MA, Khashan AS, Leahy-Warren P, Stewart F, O'Neill SM. Interventions for fear of childbirth including tocophobia. Cochrane Database Syst Rev. 2021 Jul 7;7(7):CD013321. doi: 10.1002/14651858.CD013321.pub2. PMID 34231203